CLINICAL TRIAL: NCT01491828
Title: Study to Determine Results of Vibratory Stimulus on Subject's Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kai Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 400
Record Dates: First submitted 2011-12-10; First posted 2011-12-14 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2011-12

CONDITIONS: Sleep Apnea; Snoring
Keywords: Apnea; Sleep apnea; Snoring; Hypoglossal nerve stimulation; Laynx stimulation
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Kai Strap — Medical device component that vibrates on a subject's neck.
  Other Names: Kai Patch

SUMMARY:
This study will validate whether an external vibratory stimulus applied to a subject's neck causes head, neck or jaw movement.

DETAILED DESCRIPTION:
This study will validate whether an external vibratory stimulus applied to a subject's neck causes head, neck or jaw movement, and provide information regarding the optimum location and variable vibration parameters of vibratory stimulus on a subject's neck to cause head, neck, or jaw movement. The study will also provide information whether the subject experienced or did not experience a change in sleep stage or arousal by vibratory stimulus on a subject's neck. The data gathered from this study will be used for future studies in analyzing whether such vibratory stimulus can serve as a potential treatment for sleep disorders, such as snoring and obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 18 to 80 years old
* Able to provide written informed consent for themselves and comply with study procedures.

Exclusion Criteria:

* Known hyposensitivity or hypersensitivity to vibrations on neck.
* Neurological disorder such as seizure disorder or narcolepsy.
* Psychiatric disorders currently not under control.
* Insomniacs.
* Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Head, neck, or jaw movement | 1 month
  Movement of head, neck, or jaw as evidenced by manual observation and video camera.

SECONDARY OUTCOMES:
Affect of sleep stage | 1 month
  Electrocortical arousal caused by device as measured by EEG.

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Ford Shippey III, MD, MS, Principal Investigator
Locations (1):
- Kai Medical Sleep Lab, Honolulu, Hawaii, United States